CLINICAL TRIAL: NCT06769451
Title: Radiosurgery With proTOns for the Treatment of VEntricular maLignant Tachyarrhytmias (TOVEL Study)
Brief Title: Proton Radiosurgery for the Treatment of Malignant Ventricular Tachyarrhythmias
Acronym: TOVEL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento (Other)
Collaborators: Università degli Studi di Trento (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A757
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Ventricular Arrhythmia; Ventricular Tachycardia (V-Tach)
Keywords: Stereotactic arrhythmia radioablation (STAR); Malignant ventricular Tachycardia; Ventricular Tachycardia Storm; Radiotherapy; Proton Therapy
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiosurgical ablation of a tachyarrhytmogenic substrate with Proton Therapy (Experimental): Ablation of the arrhythmogenic substrate with a single dose of 25Gy(RBE) with Proton Therapy after pretreatment diagnostics with CT, MR and electrophysiology for the definition of the arrhytmogenic substrate. Follow-up for 24 months after treatment.
  Interventions: Radiation: Stereotactic Arrhythmia Radioablation (STAR) with Proton Therapy

INTERVENTIONS:
Radiation: Stereotactic Arrhythmia Radioablation (STAR) with Proton Therapy — STAR with a single dose of 25Gy(RBE) Proton Therapy

SUMMARY:
Ventricular arrhythmias (VAs) are the leading cause of sudden cardiac death (SCD) worldwide. The implantable defibrillator (ICD) increases survival in patients at risk of VA, with data of superiority to antiarrhythmic drugs. Nevertheless, the ICD cannot prevent VAs, and shocks delivered by the device (appropriate and inappropriate) negatively impact patients' quality of life. Transcatheter ablation (TCA) is the percutaneous therapy that can eliminate VAs and prevent any recurrence. TCA is the state of the art for the treatment of drug-unresponsive VAs in patients with structural heart disease, but the prevalence of recurrence remains high (between 30% and 60%). For these reasons, several reports have recently appeared in the literature proposing a new solution for the treatment of VAs in which the use of external-beam body radiotherapy with stereotactic-radiosurgical technique (SBRT) is described. SBRT represents a rapid, noninvasive approach based on the delivery of high radiation doses of photons (25 Gy in a single fraction) to a precise location in cardiac tissue.

SBRT has entered the latest 2022 European Society of Cardiology (ESC) guidelines on VAs as a "bailout therapy". Based on preliminary data in the oncology setting, proton therapy could allow further optimization of compliance of these therapeutic doses by preserving even more of the healthy heart part and thus reducing the cardiopulmonary toxicity of radiotherapy outside the ablation target.

The investigators therefore propose an experimental (prospective interventional) study to evaluate the toxicity (primary endpoint) and efficacy (secondary endpoint) of proton radiosurgery for the treatment of VA with an enrollment of 21 patients. The primary endpoint is to evaluate the toxicity of proton radiotherapy in the acute phase (during the first 30 days of the procedure) and at 3, 6 and 12 months. A crucial part of the protocol will be the proper definition of the target to be irradiated, which will require the integration of different non-invasive cardiac imaging methodologies such as CT (Computed Tomography), MRI (Magnetic Resonance Imaging) and PET (Positron Emission Tomography), coupled with invasive and/or "non-invasive" body surface mapping with multi-electrode electrocardiogram (ECG) so as to obtain a "cardiac image" in which the myocardial scar and the arrhythmogenic region are fused.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 40 years
2. carrier of ICD/CRT-D or S-ICD
3. episodes of ventricular tachycardia/ventricular fibrillation requiring defibrillator intervention (shock or ATP) which are:

   * refractory to maximal drug therapy;
   * recurrent (at least 3 episodes in the previous 6 months);
4. patients with contraindications to a conventional ablative strategy, in relation to the high risk associated with the procedure due to the severity of the heart disease and/or the presence of comorbidities or patients who have already undergone ablation, in the presence of an arrhythmogenic substrate refractory to or unsuitable for an interventional approach or patients who refuse transcatheter ablative attempts due to high intraoperative risk in relation to the patient's characteristics.
5. Left ventricular ejection fraction ≥ 20%.

Exclusion Criteria:

1. inability to express informed consent
2. previous thoracic radiotherapy (RT) with cardiac involvement
3. active myocardial ischemia
4. recent cardiac revascularization (< 120 days)
5. hemodynamic instability (cardiogenic shock, NYHA class IV)
6. contraindication to radiosurgery (e.g., due to artifacts or other technical reasons)
7. lack of patient cooperation in pre-procedural investigations
8. ICD malfunction
9. severe comorbidity with prognosis < 12 months
10. pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Toxicity of STAR with a single dose of 25Gy(RBE) applied with Proton Therapy | Recording of MAEs for the first 24 months after therapy
  The primary endpoint will be the assessment of the toxicity of proton therapy and will be evaluated in the acute phase (during the first 30 days of the procedure) and at 3, 6, 12, 18, and 24 months. The incidence of Major Adverse Events (MAEs) related to, or presumed to be related, to proton therapy ablation will be assessed as percentage of patients with events compared to the total enrolled. The definition of MAEs (for the primary endpoint of the study) is identical to that of SAEs (as defined for reporting under Good Clinical Practice (GCP)) and can be found in the section "Serious Adverse Events (SAEs) / Major Adverse Events (MAEs) of the study protocol."

SECONDARY OUTCOMES:
Efficacy of STAR with a single dose of 25Gy(RBE) applied with Proton Therapy | Efficacy measures will be recorded for the first 24 months after therapy
  The main secondary endpoint will be the efficacy endpoint, which will involve evaluating the procedural effectiveness of therapy at 3, 6 and 12, 18 and 24 months and is the percentage reduction in VT/VF (Ventricular Tachycardia/Ventricular Fibrillation) episodes occurring after the 2-month "blanking period," compared with the period before the proton ablation procedure (6 months).
  VT episodes will be classified as follows:
  * VT episodes > 30 s, regardless of ICD intervention
  * ICD interventions on VT episodes by "antitachycardia pacing" (without shock delivery)
  * ICD interventions with appropriate DC shocks
  * Number of subjects with ≥ 50% reduction in the number of ICD treatments for VT (shock or antitachycardia pacing, ATP) comparing the 6-month period before proton therapy with the 8 months after proton therapy (excluding the 2-month blanking period after Proton Therapy).
  In addition, a series of other secondary toxicity and efficacy endpoints will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Rovereto and Proton Therapy Trento, Azienda Provinciale per i Servizi Sanitari (APSS), Trento, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zeppenfeld K, Rademaker R, Al-Ahmad A, Carbucicchio C, De Chillou C, Cvek J, Ebert M, Ho G, Kautzner J, Lambiase P, Merino JL, Lloyd M, Misra S, Pruvot E, Sapp J, Schiappacasse L, Sramko M, Stevenson WG, Zei PC, Wichterle D, Chrispin J, Siklody CH, Neuwirth R, Pelargonio G, Reichlin T, Robinson C, Tondo C. Patient selection, ventricular tachycardia substrate delineation, and data transfer for stereotactic arrhythmia radioablation: a clinical consensus statement of the European Heart Rhythm Association of the European Society of Cardiology and the Heart Rhythm Society. Europace. 2025 Mar 28;27(4):euae214. doi: 10.1093/europace/euae214. PMID 39177652
- [Background] Kovacs B, Lehmann HI, Manninger M, Saguner AM, Futyma P, Duncker D, Chun J. Stereotactic arrhythmia radioablation and its implications for modern cardiac electrophysiology: results of an EHRA survey. Europace. 2024 May 2;26(5):euae110. doi: 10.1093/europace/euae110. PMID 38666444
- [Background] Sultan A, Futyma P, Metzner A, Anic A, Richter S, Roten L, Badertscher P, Conte G, Chun JKR. Management of ventricular tachycardias: insights on centre settings, procedural workflow, endpoints, and implementation of guidelines-results from an EHRA survey. Europace. 2024 Feb 1;26(2):euae030. doi: 10.1093/europace/euae030. PMID 38363995
- [Background] Widesott L, Dionisi F, Fracchiolla F, Tommasino F, Centonze M, Amichetti M, Del Greco M. Proton or photon radiosurgery for cardiac ablation of ventricular tachycardia? Breath and ECG gated robust optimization. Phys Med. 2020 Oct;78:15-31. doi: 10.1016/j.ejmp.2020.08.021. Epub 2020 Sep 8. PMID 32911373